CLINICAL TRIAL: NCT04024163
Title: Prospective, Single-arm, Multicentre Study, Using a Historical Control, to Evaluate the Efficacy/Safety and Population Pharmacokinetics of Benznidazole in Children With Chronic Indeterminate Chagas Disease
Brief Title: Prospective Study of Benznidazole for Chagas' Disease Children With Chronic Indeterminate Chagas Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Collaborators: Chemo Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPRI747-301
Record Dates: First submitted 2019-07-14; First posted 2019-07-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Intervention Model Description: Historical control-based comparison, single-arm assignment, multicentre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Benznidazole (Experimental): Benznidazole 100 mg Tablets or Benznidazole 12.5 mg Tablets by mouth, every 12 hours for 60 days
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: Benznidazole — Drug: Benznidazole Tablets 100 mg (functionally scored) or Tablets 12.5 mg
  Other Names: National Drug Code (NDC) 0642-7464-10; National Drug Code (NDC) 0642-7464-12

SUMMARY:
This study evaluate the efficacy and safety of benznidazole in the treatment of chronic indeterminate Chagas disease in children. All subjects will receive benznidazole and results will be compared to historically to a placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 years and 18 years (age limits inclusive)
* Diagnosis of Trypanosoma cruzi (T. cruzi) infection by conventional serology based on positive ELISA and at least 1 other positive conventional serology test (recombinant ELISA or IIF)
* Written informed consent by parent/legal representative and informed assent from patients if >7 years old when applicable (as requirements may vary by country and by site)
* Females of childbearing potential (ie, female patients who have experienced menarche) and male patients must agree to use highly effective contraception if sexually active from the time of signing of the informed consent/assent form until ≥5 days after the last dose of study treatment

Exclusion Criteria:

* Pregnant or intending to become pregnant during treatment and within 5 days after the last dose of study treatment
* Patient presenting any other acute or chronic health conditions, which in the opinion of the Principal Investigator (PI), may interfere with the pharmacokinetic (PK), efficacy, and/or safety evaluation of the study treatment
* Signs and/or symptoms of acute Chagas Disease
* Known history of hypersensitivity or serious adverse reactions to nitroimidazoles
* History of Chagas Disease treatment with Benznidazole (BZN) or nifurtimox
* Immunocompromised (clinical history compatible with human immunodeficiency virus (HIV) infection, primary immunodeficiency, or prolonged treatment with corticosteroids or other immunosuppressive drugs)
* Abnormal laboratory test values (as per protocol-specified ranges) at Screening for the following parameters: total white blood cell (WBC) count, platelet count, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, and creatinine
* Abnormal ECG (as per protocol-specified ranges) and/or any Chagas disease associated findings
* Any condition that prevents the patient from taking oral medication
* Patient is known to or suspected of not being able to comply with the study protocol and the use of the investigational medicinal product (IMP)
* Evidence or history of alcohol or drug abuse (within the last 12 months)
* Any planned procedure that may interfere with highly effective contraception during treatment and within 5 days after the last dose of study treatment
* Employee of the Investigator or trial centre, or family member of the employees or the Investigator
* Any condition that, in the opinion of the Investigator, may jeopardise the trial conduct according to the protocol

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 178 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Serological Cure by Conventional ELISA | 72-month follow up
  Percentage of patients with negative conventional ELISA results as a measure of serological cure at the end of the 72-month follow up

SECONDARY OUTCOMES:
Serological Cure by Conventional ELISA at different timepoints | Day 60 (EOT), and 4, 6, 12, 24, 36, 48, 60, and 72 months of follow-up
  Percentage of patients with negative conventional ELISA results as a measure of serological cure
Serological Cure by two conventional serology tests at 72 month | 72 months of follow-up
  Percentage of patients with two negative conventional serology results as a measure of serological cure
Serological Cure by two conventional serology tests at 48 months | 48 months of follow-up
  Percentage of patients with two negative conventional serology results as a measure of serological cure
Serological Cure by three serology tests at different timepoints | Day 60 (EOT), and 4, 6, 12, 24, 36, 48, 60, and 72 months of follow-up
  Percentage of patients with three negative serology results as a measure of serological cure
Serological Cure by Non-Conventional ELISA at different timepoints | Day 60 (EOT), and 4, 6, 12, 24, 36, 48, 60, and 72 months of follow-up
  Percentage of patients with negative non-conventional ELISA (F29) results as a measure of serological cure
Cure by qPCR at different timepoints | Day 60 (EOT), and 4, 6, 12, 24, 36, 48, 60, and 72 months of follow-up
  Consistently negative quantitative polymerase chain reaction (qPCR) results as a surrogate measure of cure
Serological titres reduction at different timepoints | Day 60 (EOT), and 4, 6, 12, 24, 36, 48, 60, and 72 months of follow-up
  Reduction of conventional and nonconventional serological titres over the period of follow-up
Progression of clinical disease at different timepoints | Day 60 (EOT), and 4, 6, 12, 24, 36, 48, 60, and 72 months of follow-up
  Percentage of patients with progression to clinical disease over the period of follow-up
Progression of clinical disease and serological cure by one assay at different timepoints | 48 and 72 months of follow-up
  Percentage of patients with no evidence of established cardiomyopathy over the period of follow-up and seroconversion to negative by one assay
Progression of clinical disease and serological cure by two assays at different timepoints | 48 and 72 months of follow-up
  Percentage of patients with no evidence of established cardiomyopathy over the period of follow-up and seroconversion to negative by two assay

OTHER OUTCOMES:
Safety and Tolerability | Day 60 (EOT), and 4, 6, 12, 24, 36, 48, 60, and 72 months of follow-up
  Rate and severity of adverse events (AEs)
Population Pharmacokinetic - blood concentration | pre-dose, day 7 and day 30
  Benznidazole blood concentrations
Population Pharmacokinetic - area under the curve (AUC) | pre-dose, day 7 and day 30
  Benznidazole area under the curve (AUC)
Population Pharmacokinetic - volume of distribution | pre-dose, day 7 and day 30
  Benznidazole volume of distribution
Intensive Pharmacokinetic - blood concentrations | Day 1 or day 7
  Benznidazole blood concentrations
Intensive Pharmacokinetic - area under the curve (AUC) | Day 1 or day 7
  Benznidazole area under the curve (AUC)

CONTACTS AND LOCATIONS:
Locations (9):
- Argentina (5):
  - Hospital de Ninos "Dr. Ricardo Gutierrez", Buenos Aires
  - Hospital "Luis Carlos Lagomaggiore", Mendoza
  - Hospital Pediatrico "Dr. Humberto Notti", Mendoza
  - Hospital Público Descentralizado Dr. Guillermo Rawson, San Juan
  - Centro de Enfermedad de Chagas y Patologías Regionales, Santiago del Estero
- Bolivia (2):
  - Antigua Hospital Viedma, Cochabamba
  - CEADES - Plataforma de Chagas Sucre, Sucre
- Colombia (2):
  - Fundación Salud para el Trópico, Santa Marta
  - Centro de Atención e Investigación Médica (CAIMED), Yopal

IPD SHARING:
Plan to Share IPD: No